CLINICAL TRIAL: NCT01746641
Title: Remifentanil Versus Propofol With Target Controlled Infusion Effect Site for the Sedation of Patients During Gastrointestinal Endoscopic Procedures: Randomized Controlled Trial
Brief Title: Remifentanil Versus Propofol for TCI Sedation of Patients Undergoing Gastrointestinal Endoscopic Procedures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Occurrence of severe respiratory depression in the remifentanil group.
Sponsor: Fundación Universitaria de Ciencias de la Salud (Other)
Collaborators: Hospital de San Jose (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Acta No. 197
Record Dates: First submitted 2012-07-30; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Pain
Keywords: Remifentanil; Propofol; Sedation; Endoscopy; Gastroenterology; Target controlled infusion effect site
MeSH Terms: conditions — Pain | interventions — Remifentanil; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanil (Active Comparator): Remifentanil target controlled infusion effect site with Minto's pharmacokinetic model.
  Start dose: 1 ng/mL. Titration: 0.5 ng/mL according to clinical criteria.
  Interventions: Drug: Remifentanil
- Propofol (Active Comparator): Propofol target controlled infusion effect site with Marsh's pharmacokinetic model.
  Start dose: 1 mcg/mL. Titration: 0.5 mcg/mL according to clinical criteria.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remifentanil
  Arms: Remifentanil
Drug: Propofol
  Arms: Propofol

SUMMARY:
The purpose of this study was to compare remifentanil and propofol for sedation of patients during endoscopic gastrointestinal procedures.

DETAILED DESCRIPTION:
The administration of sedation with target controlled infusion (TCI) systems could offer a safe alternative for the management of discomfort of patients undergoing endoscopic gastrointestinal procedures. However, what medication from those available for TCI would be the most appropriate is not known.

Sixty-nine patients requiring a gastrointestinal endoscopic procedure were randomly assigned to receive a TCI effect site (e) of remifentanil (n=30) or propofol (n=39). The primary outcome was patient satisfaction. Secondary outcomes included gastroenterologist satisfaction, the proportion of adverse events between the two groups were compared (occurrence of cardiac arrhythmias, mild respiratory depression, major respiratory depression, bradycardia, hypotension, pain, nausea or vomiting, and lack of amnesia), and the level of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective higher, lower or mixed gastrointestinal endoscopy at Hospital de San Jose, Bogota, between January and December 2010.
* Be between 18 and 70 years old.
* American Society of Anesthesiology Physical Status classification between 1 and 3.
* Provide written informed consent.

Exclusion Criteria:

* Patients with difficult airway indicators.
* Pregnant women.
* Patients with chronic pain.
* Chronic opioid or benzodiazepine users (>3 months).
* Allergy history to remifentanil or propofol or eggs.
* Psychoactive drug users.
* Smokers (> 5 cigarettes per day in the previous 3 months).
* Body mass index > 30.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | At the end of the procedure, expected average of 30 minutes
  Measured with a analog scale from 1 to 4:
  1. Excellent.
  2. Good.
  3. Regular.
  4. No.

SECONDARY OUTCOMES:
Gastroenterologist satisfaction | At the end of the procedure, expected average of 30 minutes
  Measured with a analog scale from 1 to 4:
  1. Excellent.
  2. Good.
  3. Regular.
  4. No.
Adverse events | At the end of the procedure, expected average of 30 minutes
  Occurrence of cardiac arrythmias, mild respiratory depression, severe respiratory depression, bradycardia, hypotension, pain, nausea or vomiting, absence of amnesia.

OTHER OUTCOMES:
Level of consciousness | Every minute until the end of the procedure, expected average of 30 minutes
  Ramsay scale.

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Muñoz, MD, Study Director — Fundacion Universitaria de Ciencias de la Salud; Luis E Reyes, MD, Principal Investigator — Fundacion Universitaria de Ciencias de la Salud
Locations (1):
- Fundación Universitaria de Ciencias de la Salud, Bogotá, Bogota D.C., Colombia